CLINICAL TRIAL: NCT07099534
Title: Ketamine Infusion for Symptomatic Improvement in Severe Borderline Personality Disorder: A Pilot Study
Brief Title: Ketamine Infusion for Symptomatic Improvement in Severe Borderline Personality Disorder
Acronym: BorderKET
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC31/23/0619; 2024-514361-19-00 (EU CTIS Number)
Record Dates: First submitted 2025-07-25; First posted 2025-08-01 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-07

CONDITIONS: Infusion of Ketamine in Severe Borderline Personality Disorder; Borderline Personality Disorder (BPD)
Keywords: Ketamine; borderline personality disorder; BDP
MeSH Terms: conditions — Borderline Personality Disorder | interventions — Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- IV Ketamine Double Infusion (0.5 mg/kg) for Severe Borderline Personality Disorder (Experimental)
  Interventions: Drug: IV Ketamine (0.5 mg/kg) Infusion - Two Doses Administered 24 Hours Apart for Severe Borderline Personality Disorder

INTERVENTIONS:
Drug: IV Ketamine (0.5 mg/kg) Infusion - Two Doses Administered 24 Hours Apart for Severe Borderline Personality Disorder — Participants receive two intravenous (IV) infusions of ketamine at a dose of 0.5 mg/kg over 40 minutes. The first infusion is administered at Hour 0 (H0) and the second at Hour 24 (H24). Vital signs and potential adverse effects are closely monitored before, during, and after each infusion. This intervention aims to assess the short-term efficacy and safety of ketamine in reducing symptoms of severe borderline personality disorder.

SUMMARY:
The main objective of this pilot study is to evaluate at D9 the evolution of BPD symptoms' intensity(scale BSL-23) in severe BPD patients, after two Ketamine infusions (0.5mg/kg at H0 and H24). The intervention is combined with the first level standard of care : Good Psychiatric Management (GPM). Patients are followed up to 3 months by regular visits conducted by a psychiatrist. Secondary outcomes are monitored including BPD symptoms at different times, suicidal ideation, depressiv symptoms, healthcare use and adverse effects.

DETAILED DESCRIPTION:
Borderline personality disorder is a burden for patient's life and remains undertreated, no medication has FDA or AMM approval for this indication. On a neurobiological level, BPD is thought to involve defects in the regulation of the glutamatergic pathway, as well as circuit anomalies in the emotional pathways (limbic hyperactivation and deficient activation of the prefrontal cortex), which have been associated with impulsivity and emotional hyper-reactivity. Ketamine, an NMDA antagonist, has a pharmacological profile of interest for TPB, thanks to its excitatory action on the CPF and its inhibitory effect on limbic hyperactivity. Preliminary clinical data suggest an effect on TPB symptomatology, more data is needed to conduct a large scale study.

This pilot study aim to test the effect of two infusions of ketamine (0,5 mg/kg) in adults with severe BPD. The protocol consists of two IV ketamine injections over 40 min at a dose of 0.5 mg/kg each, at H0 and H24.The associated treatment will be in line with first-level recommendations, i.e. GPM-type psychotherapy.

Infusions are delivered under medical monitoring at hospital and patients are followed up to 3 months by regular psychiatric consultations. Change in BPD symptoms'intensity is measured by the scale BSL-23 at different times (baseline, H48, J9, J28, M3) up to 3 months. Suicidal ideations, depressive symptoms, health care sue and adverse effects are also monitored.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient aged 18 to 65 years
* Fluent in French
* Person affiliated with or receiving social security benefits.
* Diagnosis of borderline personality disorder established according to the DSM-5 MINI criteria (5 out of 9 criteria)
* Severe borderline personality disorder
* Patient receiving stable pharmacological (antipsychotic, mood stabilizer, antidepressant) and/or non-pharmacological (schema therapy, DBT) treatment for four weeks

Exclusion Criteria:

* Personal history of an acute psychotic episode or chronic psychotic disorder
* Personal history of a manic or hypomanic episode
* Family history (first-degree relatives) of a psychotic disorder
* Current severe depressive episode
* Recreational ketamine use (multi-weekly ketamine use)
* New long-term treatment introduced within the previous four weeks (antidepressant, antipsychotic, mood stabilizer)
* Prescription of an Monoamine oxidase inhibitors (increased risk of hypertension)
* Specific absolute contraindication to ketamine
* History of cirrhosis or major liver function test abnormalities
* Major ECG abnormality

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Borderline Personality Disorder Symptom Severity (BSL-23) from Baseline (H0) to Day 9 (J9) | Baseline and Day 9 post perfusion
  The primary outcome measure is the change in symptom severity of Borderline Personality Disorder (BPD) as assessed by the Borderline Symptom List-23 (BSL-23) from Baseline to Day 9 post perfusion. The BSL-23 is a self-reported scale measuring BPD symptom intensity, with scores ranging from 0 (no symptoms) to 92 (most severe symptoms). A higher score indicates greater symptom severity. The difference in total BSL-23 scores between Baseline and Day 9 will be analyzed to evaluate the short-term impact of IV ketamine treatment on BPD symptoms.

SECONDARY OUTCOMES:
Change in Borderline Personality Disorder Symptom Severity (BSL-23) from Baseline to H48, Month 1 (M1), and Month 3 (M3) | Baseline, 48 hours, 1 month, and 3 months after first ketamine infusion.
  This secondary outcome measure evaluates changes in symptom severity of Borderline Personality Disorder (BPD) using the Borderline Symptom List-23 (BSL-23) at multiple time points: H48, Month 1 (M1), and Month 3 (M3), compared to Baseline. The BSL-23 is a self-reported scale assessing BPD symptoms, with total scores ranging from 0 (no symptoms) to 92 (most severe symptoms). Higher scores indicate greater symptom severity. The difference in scores across these time points will be analyzed to assess the medium- to long-term impact of IV ketamine treatment on BPD symptoms.
Change in Borderline Personality Disorder Symptom Severity Measured by Zanarini-BPD Scale from Baseline to H48, D9, M1, and M3 | Baseline, 48 hours, Day 9, 1 month, and 3 months after first ketamine infusion.
  The Zanarini-BPD scale assesses the severity of borderline personality disorder symptoms based on nine DSM-IV criteria. Each criterion is rated on a Likert scale from 0 to 4, with higher scores indicating greater symptom severity. The total score ranges from 0 to 36. This outcome measures the change in symptom severity from baseline to H48, D9, M1, and M3.
Change in Suicidal Ideation Severity Measured by C-SSRS from Baseline to H48, D9, M1, and M3 | Baseline, 48 hours, Day 9, 1 month, and 3 months after first ketamine infusion.
  The Columbia-Suicide Severity Rating Scale (C-SSRS) assesses suicidal ideation severity based on structured interview questions. Scores range from 0 (no suicidal ideation) to 5 (active suicidal intent with a plan). This outcome measures changes in severity from baseline to H48, D9, M1, and M3.
Change in Depressive Symptom Severity Measured by MADRS from Baseline to H48, D9, M1, and M3 | Baseline, 48 hours, Day 9, 1 month, and 3 months after first ketamine infusion.
  The Montgomery-Åsberg Depression Rating Scale (MADRS) assesses the severity of depressive symptoms based on a structured clinical interview. The scale includes 10 items, each rated from 0 (no symptoms) to 6 (severe symptoms), with a total score ranging from 0 to 60. Higher scores indicate more severe depression. This outcome measures changes in depressive symptom severity from baseline to H48, D9, M1, and M3.
Number of Psychiatric Emergency Room Visits (Self-Reported, Day 9 to Month 3) | From Day 9 (J9) to Month 3 (M3)
  This outcome measure tracks the number of psychiatric emergency room visits reported by participants between Day 9 (J9) and Month 3 (M3). Visits are self-reported during follow-up assessments and, when possible, cross-checked with medical records. A psychiatric emergency visit is defined as any unplanned presentation to an emergency department for acute psychiatric symptoms, crisis management, or safety concerns. The data will be analyzed to evaluate the impact of IV ketamine treatment on emergency psychiatric care utilization over time.

CONTACTS AND LOCATIONS:
Locations (1):
- Toulouse Purpan University Hospital, Head of Psychiatry Clinic in the UF3 department, Toulouse, France

IPD SHARING:
Plan to Share IPD: No